CLINICAL TRIAL: NCT02460692
Title: A Randomized Controlled Trial of Dronabinol and Vaporized Cannabis in Chronic Low Back Pain
Brief Title: Trial of Dronabinol and Vaporized Cannabis in Chronic Low Back Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Thomas D. Marcotte, PhD, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1R01DA038634-01A1 (NIH); R01DA038634 (NIH)
Record Dates: First submitted 2015-05-29; First posted 2015-06-02 (Estimated); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Cannabis; Low Back Pain; Neuropathic Pain
MeSH Terms: conditions — Marijuana Abuse; Low Back Pain; Neuralgia | interventions — Sugars; Dronabinol; nabiximols

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebos (Placebo Comparator): The present study is designed to evaluate whether or not a medium dose of cannabis (3.7% delta-9-THC/5.6% CBD) can maintain an analgesic response over an eight week period compared to placebo.
  Interventions: Drug: Placebos
- Dronabinol (Active Comparator): A direct comparison of cannabis and dronabinol has not been performed in a clinical population. The present study will fill this void by performing a randomized, controlled 8 week trial comparing the effectiveness of oral versus vaporized cannabis in patients with neuropathic low back pain.
  Interventions: Drug: dronabinol
- Vaporized Cannabis 3.7% THC/5.6% CBD (Experimental): The eight week outpatient study will compare the efficacy and side effect profile of cannabis (3.7%THC/5.6%CBD) and dronabinol. We will also perform a human laboratory experiment evaluating driving using the same study medications that subjects received during their 8 week outpatient treatment.
  Interventions: Drug: Vaporized Cannabis 3.7% THC/5.6% CBD

INTERVENTIONS:
Drug: Placebos — Administration of vaporized cannabis plus either dronabinol or placebo pill
  Other Names: sugar pill
  Arms: Placebos
Drug: dronabinol — Administration of vaporized cannabis plus either dronabinol or placebo pill
  Other Names: Marinol
  Arms: Dronabinol
Drug: Vaporized Cannabis 3.7% THC/5.6% CBD — Administration of vaporized cannabis plus either dronabinol or placebo pill
  Other Names: marijuana
  Arms: Vaporized Cannabis 3.7% THC/5.6% CBD

SUMMARY:
This study will involve treating low back pain associated with nerve injury with oral delta-9-tetrahydrocannabinol (Δ9-THC) or whole plant cannabis for eight weeks. Research subjects will consume either oral Δ9-THC (dronabinol), vaporized 3.7% Δ9-THC/5.6% CBD, or placebo. An analysis will then be determined to assess the risk--benefit ratio of dronabinol and vaporized 3.7% Δ9-THC/5.6% CBD .

DETAILED DESCRIPTION:
The present study is designed to assess whether treatment with vaporized cannabis or dronabinol (oral Δ9-THC) reduces spontaneous and evoked pain more than placebo, and whether there are any differences between the two active treatments in terms of interference with activities of daily living. This study also aims to examine the effects of vaporized whole plant cannabis and dronabinol on mood, neuropsychological function, and psychomimetic side-effects (high, stoned, etc.) compared to placebo and to each other. In addition, we plan to examine the acute effects (after receiving stable treatment for 4 weeks) of vaporized cannabis and dronabinol compared to placebo and each other on driving skills.

ELIGIBILITY:
Inclusion Criteria:

Age greater than 18. Presence of chronic low back pain (CLBP) defined as the response to two questions 1) How long has back pain been an ongoing problem for you? 2) How often has low back pain been an ongoing problem for you over the past 6 months? A response of greater than 3 months to question 1 and a response of "at least half the days in the past 6 months" to question 2 will define CLBP according to the NIH Task Force on Research Standards for Chronic Low Back Pain.

The numerical pain intensity must be greater than 3/10 each day during the one-week observation period.

To avoid confounding by concurrent medications, participants will have had a stable analgesic regimen that they will continue throughout the study To obviate residual neuropsychological effects from cannabis exposure, participants will be abstinent from this herbal medicine for 7 days prior to study entry.

Exclusion Criteria:

Presence of another painful condition of greater severity than the neuropathic pain condition which is being studied.

History of traumatic brain injury. Clinically significant or unstable medical condition. Individuals with significant cardiovascular, hepatic or renal disease, uncontrolled hypertension, and chronic pulmonary disease (eg, asthma, COPD), will be excluded. If warranted clinically, subjects will undergo laboratory evaluation (blood chemistry, electrocardiogram, urinalysis, toxicology screening for confirmation. Females of childbearing potential will undergo pregnancy testing.

A positive result on toxicity screening will exclude individuals from participation. A urine drug test that screens for 5 categories of drugs: marijuana (Δ9-THC), cocaine, amphetamines/methamphetamines, opiates, benzodiazepines and phencyclidine (PCP) will be employed. A positive result for opioids and/or THC will not be exclusionary if the patient is receiving a prescription for an opioid and/or THC.

Allergy to sesame oil, lactose, or gelatin Vascular disease, especially Raynauld's syndrome, systolic blood pressure > 170 mm, diastolic blood pressure > 100 mm Recent injuries to the upper extremity Cognitive impairment, such as Dementia or Alzheimer's Disease Substance Abuse History: The Substance Abuse Module of the Diagnostic Interview Schedule for the Diagnostic and Statistical Manual (DSM)-IV will be administered to exclude individuals with current substance use disorders.

Pregnancy as ascertained by a mandatory commercial pregnancy test Past history of suicide attempt. Cannabis can exacerbate pre-existing schizophrenia, and has been linked to an increase in the risk of suicide in such patients. In patients with bipolar disorder, cannabis use has been associated with worsening of manic and psychotic symptoms. Such findings suggest that cannabis is contraindicated in individuals with serious mental health issues, a line of reasoning that will be observed in the present study by excluding patients in the bipolar/schizoaffective/schizophrenic spectrum.

Suicidality. Exposure to cannabis does not lead to depression but it may be associated with suicidal thoughts and attempts. Therefore, the Beck Depression Inventory (BDI)-II will be used to measure suicidal ideation.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2020-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas D Marcotte, PhD, Principal Investigator — UC San Diego
Locations (1):
- UC Center for Medicinal Cannabis Research, UC San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wilsey B, Marcotte T, Tsodikov A, Millman J, Bentley H, Gouaux B, Fishman S. A randomized, placebo-controlled, crossover trial of cannabis cigarettes in neuropathic pain. J Pain. 2008 Jun;9(6):506-21. doi: 10.1016/j.jpain.2007.12.010. Epub 2008 Apr 10. PMID 18403272
- [Background] Wilsey B, Marcotte T, Deutsch R, Gouaux B, Sakai S, Donaghe H. Low-dose vaporized cannabis significantly improves neuropathic pain. J Pain. 2013 Feb;14(2):136-48. doi: 10.1016/j.jpain.2012.10.009. Epub 2012 Dec 11. PMID 23237736
- [Background] Wilsey B, Atkinson JH, Marcotte TD, Grant I. The Medicinal Cannabis Treatment Agreement: Providing Information to Chronic Pain Patients Through a Written Document. Clin J Pain. 2015 Dec;31(12):1087-96. doi: 10.1097/AJP.0000000000000145. PMID 25370134
- [Background] Grant I, Atkinson JH, Gouaux B, Wilsey B. Medical marijuana: clearing away the smoke. Open Neurol J. 2012;6:18-25. doi: 10.2174/1874205X01206010018. Epub 2012 May 4. PMID 22629287

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebos: The present study is designed to evaluate whether or not a medium dose of cannabis (3.7% delta-9-Tetrahydrocannabinol (THC)/5.6% CBD) can maintain an analgesic response over an eight week period compared to placebo.
  Placebos: Administration of vaporized cannabis plus either dronabinol or placebo pill
  During the titration period (weeks 0-4), participants undergo titration of vaporized medication from 4 puffs to 18 puffs, or oral medication from 5 mg qd to 10 mg tid per day. During the treatment period (weeks 5-8), participants are expected to consume the amount of study medication that they titrated themselves up to by the end of week 4.
- Dronabinol: A direct comparison of cannabis and dronabinol has not been performed in a clinical population. The present study will fill this void by performing a randomized, controlled 8 week trial comparing the effectiveness of oral versus vaporized cannabis in patients with neuropathic low back pain.
  dronabinol: Administration of vaporized cannabis plus either dronabinol or placebo pill
  During the titration period (weeks 0-4), participants undergo titration of vaporized medication from 4 puffs to 18 puffs, or oral medication from 5 mg qd to 10 mg tid per day. During the treatment period (weeks 5-8), participants are expected to consume the amount of study medication that they titrated themselves up to by the end of week 4
- Vaporized Cannabis 3.7% THC/5.6% CBD: The eight week outpatient study will compare the efficacy and side effect profile of cannabis (3.7%THC/5.6%CBD) and dronabinol. We will also perform a human laboratory experiment evaluating driving using the same study medications that subjects received during their 8 week outpatient treatment.
  Vaporized Cannabis 3.7% THC/5.6% CBD: Administration of vaporized cannabis plus either dronabinol or placebo pill
  During the titration period (weeks 0-4), participants undergo titration of vaporized medication from 4 puffs to 18 puffs, or oral medication from 5 mg qd to 10 mg tid per day. During the treatment period (weeks 5-8), participants are expected to consume the amount of study medication that they titrated themselves up to by the end of week 4
Period: Overall Study
Arm/Group | Placebos | Dronabinol | Vaporized Cannabis 3.7% THC/5.6% CBD
Started | 44 | 43 | 44
Completed | 29 | 26 | 36
Not Completed | 15 | 17 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebos | Dronabinol | Vaporized Cannabis 3.7% THC/5.6% CBD | Total
Number analyzed (Participants) | 44 | 43 | 44 | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.8 (13.7) | 48.6 (13) | 47.4 (12.3) | 44.9 (13.6)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 21 | 20 | 20 | 61
  Gender: Male | 23 | 21 | 23 | 67
  Gender: Transgender (Female to Male) | 0 | 1 | 0 | 1
  Gender: Transgender (Male to Female) | 0 | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 10 | 8 | 29
  Not Hispanic or Latino | 33 | 33 | 36 | 102
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2 | 4
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 7 | 10 | 7 | 24
  White | 27 | 22 | 29 | 78
  More than one race | 4 | 3 | 4 | 11
  Unknown or Not Reported | 4 | 6 | 1 | 11
Education [Mean (Standard Deviation); unit: Years] | 14.2 (2.2) | 13.8 (2.4) | 14.6 (2.6) | 14.2 (2.39)

OUTCOME MEASURES:

1. Primary Outcome: Numerical Pain Intensity
Description: The primary outcome is self-reported daily average numerical pain intensity during the past 24 hours. The numerical pain intensity is an 11-point pain intensity numerical rating scale (PI-NRS), where 0 equals no pain and 10 equals worst possible pain. The time frame includes baseline and weeks 1, 3, 5, 7, 8. Baseline is the pain tensity reported at the first day in the daily diary, before the first dose. The follow-up pain intensities (weeks 1, 3, 5, 7, 8) are the daily diary average pain intensities since the previously reported timepoint.
Time Frame: 8 weeks
Population: There are missing values.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebos | Dronabinol | Vaporized Cannabis 3.7% THC/5.6% CBD
Number analyzed (Participants) | 39 | 37 | 41
score on a scale
  Baseline | 6.03 (1.65) | 6.11 (1.65) | 6.24 (1.87)
  Week 1: number analyzed (Participants) | 36 | 36 | 41
  Week 1 | 5.97 (2.01) | 5.80 (1.62) | 5.64 (1.98)
  Week 3: number analyzed (Participants) | 32 | 35 | 40
  Week 3 | 5.65 (1.56) | 5.67 (1.62) | 5.43 (2.11)
  Week 5: number analyzed (Participants) | 29 | 30 | 36
  Week 5 | 5.47 (1.77) | 4.89 (1.88) | 4.82 (2.29)
  Week 7: number analyzed (Participants) | 26 | 28 | 34
  Week 7 | 5.26 (1.80) | 4.35 (2.02) | 4.72 (2.23)
  Week 8: number analyzed (Participants) | 26 | 26 | 33
  Week 8 | 5.22 (1.92) | 4.19 (2.02) | 4.45 (2.11)
Statistical Analysis 1: Comparison: Dronabinol vs Vaporized Cannabis 3.7% THC/5.6% CBD; This is the primary comparison; Test type: Superiority; p = 0.78, unstructured covariance model — The average pain change at the treatment period (weeks 5-8) from baseline were compared between the two arms using an unstructured covariance model, excluding main group effect
Statistical Analysis 2: Comparison: Placebos vs Vaporized Cannabis 3.7% THC/5.6% CBD; This is the secondary comparison; Test type: Superiority; p = 0.070, Unstructured covariance model — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebos vs Dronabinol; This is an exploratory comparison; Test type: Superiority; p = 0.044, Unstructured covariance model — [p-value comment as in outcome 1, analysis 1]

2. Secondary Outcome: Repeated Measures Recommended Minimal Dataset (NIH Task Force on Chronic Low Back Pain)
Description: A Task Force was convened by the NIH Pain Consortium, with the goal of developing research standards for chronic low back pain. The results included recommendations for a repeated measures dataset in order to establish greater consistency in reporting in order to facilitate comparisons among studies. The repeated measure minimal dataset is based upon scores based upon the Patient-Reported Outcomes Measurement Information System ® (PROMIS). These items yield a classification of impacts on the lives of patients that range from 1 (least impact) to 42 (greatest impact).
Time Frame: 8 weeks
Population: There were some missing data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebos | Dronabinol | Vaporized Cannabis 3.7% THC/5.6% CBD
Number analyzed (Participants) | 44 | 42 | 44
score on a scale
  Baseline | 21.6 (7.29) | 22.5 (6.46) | 23.1 (7.03)
  Week 1: number analyzed (Participants) | 37 | 37 | 41
  Week 1 | 18.5 (8.97) | 19.9 (6.48) | 20.3 (8.08)
  Week 3: number analyzed (Participants) | 29 | 34 | 39
  Week 3 | 17.2 (7.40) | 18.1 (7.44) | 19.2 (9.30)
  Week 5: number analyzed (Participants) | 28 | 31 | 36
  Week 5 | 16.3 (7.70) | 16.9 (6.93) | 16.6 (9.18)
  Week 7: number analyzed (Participants) | 28 | 28 | 35
  Week 7 | 16.2 (7.42) | 15.1 (7.17) | 16.1 (9.88)
  Week 8: number analyzed (Participants) | 28 | 28 | 36
  Week 8 | 15.9 (9.06) | 15.8 (8.53) | 15.8 (10.3)
Statistical Analysis 1: Comparison: Dronabinol vs Vaporized Cannabis 3.7% THC/5.6% CBD; Test type: Superiority; p = 0.27, unstructured covariance model — The average change of impact scores at the treatment period (weeks 5-8) from baseline were compared between the two arms using an unstructured covariance model, excluding main group effect
Statistical Analysis 2: Comparison: Placebos vs Dronabinol; Test type: Superiority; p = 0.96, unstructured covariance model — The average change of impact scores at the treatment period (weeks 5-8) from baseline were compared between the arms using an unstructured covariance model, excluding main group effect
Statistical Analysis 3: Comparison: Placebos vs Vaporized Cannabis 3.7% THC/5.6% CBD; Test type: Superiority; p = 0.30, unstructured covariance model — [p-value comment as in outcome 2, analysis 1]

3. Secondary Outcome: Neuropathic Pain Scale
Description: The Neuropathic Pain Scale (NPS) is an 11-point numerical scale consisting of 13 questions that ask ratings of various pain descriptors (including pain intensity, sharpness, burning, aching, cold, sensitivity, itching,unpleasantness, deep, and surface pain). The NPS is scored as the sum of these pain descriptors. Range of scores is from 0 to100. A higher score is a worse score.
Time Frame: 8 weeks
Population: Some subjects dropped out before completing the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebos | Dronabinol | Vaporized Cannabis 3.7% THC/5.6% CBD
Number analyzed (Participants) | 44 | 43 | 44
score on a scale
  Baseline: number analyzed (Participants) | 43 | 42 | 43
  Baseline | 45.9 (15.2) | 45.1 (13.5) | 48.3 (15.7)
  Week 1: number analyzed (Participants) | 37 | 36 | 41
  Week 1 | 40.4 (16.7) | 38.9 (12.0) | 42.3 (15.9)
  Week 3: number analyzed (Participants) | 29 | 34 | 39
  Week 3 | 37.0 (17.2) | 34.6 (13.6) | 39.2 (19.1)
  Week 5: number analyzed (Participants) | 28 | 29 | 36
  Week 5 | 35.1 (16.4) | 30.8 (14.8) | 37.5 (17.6)
  Week 7: number analyzed (Participants) | 28 | 28 | 35
  Week 7 | 36.0 (17.8) | 29.6 (14.8) | 33.4 (19.7)
  Week 8: number analyzed (Participants) | 28 | 27 | 36
  Week 8 | 34.6 (18.3) | 28.2 (16.3) | 33.2 (20.4)
Statistical Analysis 1: Comparison: Dronabinol vs Vaporized Cannabis 3.7% THC/5.6% CBD; Test type: Superiority; p = 0.44, unstructured covariance model — The average NPS change at the treatment period (weeks 5-8) from baseline were compared between the two arms using an unstructured covariance model, excluding main group effect
Statistical Analysis 2: Comparison: Placebos vs Vaporized Cannabis 3.7% THC/5.6% CBD; Test type: Superiority; p = 0.53, Unstructured covariance model — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebos vs Dronabinol; Test type: Superiority; p = 0.18, Unstructured covariance model — [p-value comment as in outcome 3, analysis 1]

4. Secondary Outcome: Hopkins Verbal Learning Test
Description: The Hopkins Verbal Learning Test provides information on the ability to learn and immediately recall verbal information across trials, as well at the ability to retain, reproduce, and recognize this information after a delay. A list of 12 words is presented to the subject over three trials. After each trial, the subject is to recall as many items as possible from the list in any desired order. A 20-minute delay follows the administration of the three trials, after which the subject is asked to recall the list.
  The ability to learn is represented by the number of correct words, with a score range of 0-36. A higher score indicates better performance.
Time Frame: 8 weeks
Population: Some subjects dropped out before completing the study.
Measure: Mean (Standard Deviation); unit: Number of correct words
Arm/Group | Placebos | Dronabinol | Vaporized Cannabis 3.7% THC/5.6% CBD
Number analyzed (Participants) | 44 | 42 | 44
Number of correct words
  Baseline | 24.1 (5.24) | 23.7 (5.21) | 24.4 (4.90)
  Week 1: number analyzed (Participants) | 35 | 35 | 42
  Week 1 | 24.0 (4.78) | 23.3 (4.44) | 24.0 (4.44)
  Week 3: number analyzed (Participants) | 29 | 32 | 39
  Week 3 | 22.9 (3.74) | 23.6 (5.04) | 22.8 (4.08)
  Week 5: number analyzed (Participants) | 29 | 28 | 36
  Week 5 | 25.6 (3.84) | 24.0 (4.90) | 24.6 (4.55)
  Week 7: number analyzed (Participants) | 28 | 28 | 35
  Week 7 | 24.3 (4.00) | 24.7 (4.78) | 23.8 (4.99)
  Week 8: number analyzed (Participants) | 28 | 28 | 35
  Week 8 | 24.0 (4.16) | 24.5 (4.68) | 24.8 (5.53)
Statistical Analysis 1: Comparison: Dronabinol vs Vaporized Cannabis 3.7% THC/5.6% CBD; Test type: Superiority; p = 0.95, unstructured covariance model — The average change of learning scores at the treatment period (weeks 5-8) from baseline were compared between the arms using an unstructured covariance model, excluding main group effect
Statistical Analysis 2: Comparison: Placebos vs Vaporized Cannabis 3.7% THC/5.6% CBD; Test type: Superiority; p = 0.94, unstructured covariance model — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Placebos vs Dronabinol; Test type: Superiority; p = .90, unstructured covariance model — The average change of learning score at the treatment period (weeks 5-8) from baseline were compared between the arms using an unstructured covariance model, excluding main group effect

5. Secondary Outcome: Grooved Pegboard Test - Dominant Hand
Description: The Grooved Pegboard Test is a test of fine motor coordination and speed. Subjects are required to place 25 small metal pegs into holes on a 3" x 3" metal board. All pegs are alike and have a ridge on one side, which corresponds to a notch in each hole on the board. First the dominant hand is tested, and subjects are asked to place the pegs in the holes as fast as they can. This is then repeated with the non-dominant hand, and the total time for each hand is recorded. A higher score indicates worse performance.
Time Frame: 8 weeks
Population: There were some missing data.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Placebos | Dronabinol | Vaporized Cannabis 3.7% THC/5.6% CBD
Number analyzed (Participants) | 44 | 42 | 43
seconds
  Baseline | 63.7 (10.6) | 73.4 (21.1) | 69.1 (14.4)
  Week 1: number analyzed (Participants) | 35 | 35 | 41
  Week 1 | 60.7 (9.83) | 69.5 (23.8) | 64.5 (13.2)
  Week 3: number analyzed (Participants) | 28 | 31 | 39
  Week 3 | 61.1 (14.1) | 63.1 (10.9) | 64.1 (11.2)
  Week 5: number analyzed (Participants) | 26 | 28 | 35
  Week 5 | 59.9 (14.8) | 69.0 (23.3) | 61.7 (12.1)
  Week 7: number analyzed (Participants) | 27 | 27 | 35
  Week 7 | 59.7 (13.6) | 68.7 (24.9) | 62.5 (13.3)
  Week 8: number analyzed (Participants) | 28 | 27 | 35
  Week 8 | 60.8 (18.5) | 69.2 (27.6) | 61.7 (12.7)
Statistical Analysis 1: Comparison: Dronabinol vs Vaporized Cannabis 3.7% THC/5.6% CBD; Test type: Superiority; p = 0.93, unstructured covariance model — The average change of total time completing task in grooved pegboard test on dominant hand (weeks 5-8 at the treatment period) from baseline were compared between the two arms using an unstructured covariance model
Statistical Analysis 2: Comparison: Placebos vs Dronabinol; Test type: Superiority; p = 0.92, unstructured covariance model — The average change of total time completing task in grooved pegboard test on dominant hand (weeks 5-8, at the treatment period) from baseline were compared between the two arms using an unstructured covariance model
Statistical Analysis 3: Comparison: Placebos vs Vaporized Cannabis 3.7% THC/5.6% CBD; Test type: Superiority; p = 0.85, unstructured covariance model — [p-value comment as in outcome 5, analysis 2]

6. Secondary Outcome: Wechsler Adult Intelligence Scale-III Digit Symbol Test
Description: The Digit Symbol test measures concentration, psychomotor speed, and graphomotor abilities. This pen and paper test involves having subjects substitute a series of symbols with numbers as quickly and accurately as possible during a 120 second period. The results are expressed as the number of correct substitutions with a score range of 0-133. A higher number indicates better performance.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: number of correct symbols
Arm/Group | Placebos | Dronabinol | Vaporized Cannabis 3.7% THC/5.6% CBD
Number analyzed (Participants) | 44 | 43 | 42
number of correct symbols
  Baseline | 80.3 (14.9) | 69.6 (17.2) | 72.2 (15.6)
  Week 1 | 84.8 (17.2) | 73.5 (19.3) | 78.3 (16.7)
  Week 3 | 88.9 (17.5) | 75.6 (18.2) | 77.6 (19.7)
  Week 5 | 90.0 (19.7) | 79.2 (20.9) | 83.1 (18.8)
  Week 7 | 88.4 (20.9) | 79.8 (19.8) | 81.0 (21.3)
  Week 8 | 84.8 (22.6) | 79.3 (21.9) | 87.3 (18.6)
Statistical Analysis 1: Comparison: Dronabinol vs Vaporized Cannabis 3.7% THC/5.6% CBD; Test type: Superiority; p = 0.89, Unstructured covariance model — The average change in Wechsler Adult Intelligence Scale (WAIS)-III test score (weeks 5-8, at the treatment period) from baseline were compared between the two arms using an unstructured covariance model
Statistical Analysis 2: Comparison: Placebos vs Dronabinol; Test type: Superiority; p = 0.13, unstructured covariance model — The average change in WAIS-III test score (weeks 5-8, at the treatment period) from baseline were compared between the two arms using an unstructured covariance model
Statistical Analysis 3: Comparison: Placebos vs Vaporized Cannabis 3.7% THC/5.6% CBD; Test type: Superiority; p = 0.14, unstructured covariance model — [p-value comment as in outcome 6, analysis 2]

7. Secondary Outcome: Profile of Mood States
Description: This questionnaire contains 65 words/statements that describe feelings people have. The questionnaire requires the patient to indicate for each word or statement how he or she has been feeling in the past week. There are 6 subscales: tension-anxiety (9 items, score range: 0-36), depression (15 items, range 0-60), anger-hostility (12 items, range 0-48), vigor-activity (8 items, range 0-32), fatigue (7 items, range 0-28), confusion-bewilderment (7 items, range 0-28).
  The total mood disturbance (TMD) is calculated by adding the scores for tension-anxiety, depression, anger-hostility, fatigue and confusion-bewilderment and then subtracting the score for vigor-activity. The TMD is reported and has a score range of -32 to 200. A higher score indicates worse symptoms.
Time Frame: 8 weeks
Population: There were some missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebos | Dronabinol | Vaporized Cannabis 3.7% THC/5.6% CBD
Number analyzed (Participants) | 44 | 42 | 44
score on a scale
  Baseline | 57.3 (32.0) | 53.8 (31.5) | 53.2 (30.6)
  Week 1: number analyzed (Participants) | 37 | 36 | 44
  Week 1 | 51.5 (36.9) | 46.2 (23.6) | 41.5 (22.2)
  Week 3: number analyzed (Participants) | 29 | 34 | 39
  Week 3 | 48.6 (30.6) | 42.9 (27.4) | 38.8 (23.3)
  Week 5: number analyzed (Participants) | 28 | 29 | 35
  Week 5 | 46.3 (27.2) | 40.0 (22.7) | 38.8 (22.0)
  Week 7: number analyzed (Participants) | 28 | 28 | 35
  Week 7 | 45.5 (27.3) | 37.7 (23.7) | 44.2 (29.2)
  Week 8: number analyzed (Participants) | 27 | 28 | 35
  Week 8 | 42.5 (30.9) | 41.0 (28.5) | 39.7 (26.6)
Statistical Analysis 1: Comparison: Dronabinol vs Vaporized Cannabis 3.7% THC/5.6% CBD; Test type: Superiority; p = 0.10, Unstructured covariance model — The average change of total mood disturbance scores (weeks 5-8, at the treatment period) from baseline were compared between the two arms using an unstructured covariance model, excluding main group effect
Statistical Analysis 2: Comparison: Placebos vs Dronabinol; Test type: Superiority; p = 0.67, unstructured covariance model — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 3: Comparison: Placebos vs Vaporized Cannabis 3.7% THC/5.6% CBD; Test type: Superiority; p = 0.25, unstructured covariance model — [p-value comment as in outcome 7, analysis 1]

8. Secondary Outcome: Beck Depression Inventory II
Description: The Beck Depression Inventory is composed of items relating to symptoms of depression such as hopelessness and irritability, cognitions such as guilt or feelings of being punished, as well as physical symptoms such as fatigue, weight loss, and lack of interest in sex. Range of scores is from 0 to 63. A higher score is a worse score.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebos | Dronabinol | Vaporized Cannabis 3.7% THC/5.6% CBD
Number analyzed (Participants) | 41 | 42 | 44
score on a scale
  Baseline | 8.05 (7.99) | 7.81 (8.26) | 7.84 (8.14)
  Week 1 | 7.68 (8.70) | 5.61 (5.00) | 5.32 (6.05)
  Week 3 | 5.76 (6.59) | 5.26 (6.81) | 5.59 (7.24)
  Week 5 | 5.32 (7.07) | 5.52 (6.28) | 6.25 (8.52)
  Week 7 | 5.50 (7.63) | 4.36 (6.49) | 6.09 (8.63)
  Week 8 | 5.32 (7.39) | 5.25 (8.11) | 6.06 (9.62)
Statistical Analysis 1: Comparison: Dronabinol vs Vaporized Cannabis 3.7% THC/5.6% CBD; Test type: Superiority; p = 0.84, unstructured covariance model — The average change of beck score (weeks 5-8 at the treatment period) from baseline were compared between the arms using an unstructured covariance model, excluding main group effect
Statistical Analysis 2: Comparison: Placebos vs Dronabinol; Test type: Superiority; p = 0.91, unstructured covariance model — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Placebos vs Vaporized Cannabis 3.7% THC/5.6% CBD; Test type: Superiority; p = 0.75, unstructured covariance model — [p-value comment as in outcome 8, analysis 1]

9. Secondary Outcome: Locally Developed Psychoactive Effect Scale - Good Drug Effect
Description: Visual Analogue Scale (VAS) ratings will be presented as a 100-mm horizontal line, anchored on the left with 'not at all' and on the right with 'extremely'. Participants will pencil in a vertical line along the horizontal line that represents their current feeling (questions usually phrased, 'During the past week, did you feel ___after consuming the vaporized cannabis?'). Ratings will be: any drug effect, a good drug effect, a bad drug effect, high, drunk, impaired, stoned, as if you liked the drug effect, sedated, confused, nauseous, like you desired more of the drug, anxious, down, and very hungry.
  This is a substudy. A good drug effect is presented. Range of scores is from 0 to 100. A higher score is a worse score.
Time Frame: 6 hours
Population: There are some missing values
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebos | Dronabinol | Vaporized Cannabis 3.7% THC/5.6% CBD
Number analyzed (Participants) | 8 | 13 | 21
score on a scale
  After dose 1 hour: number analyzed (Participants) | 8 | 13 | 20
  After dose 1 hour | 14.2 (24.4) | 19.1 (34.3) | 58.8 (32.5)
  After dose 2 hours | 14.0 (23.8) | 33.5 (38.5) | 45.7 (31.7)
  After dose 3 hours: number analyzed (Participants) | 8 | 12 | 21
  After dose 3 hours | 5.88 (14.3) | 33.2 (44.1) | 27.5 (29.5)
  After dose 4 hours: number analyzed (Participants) | 7 | 13 | 21
  After dose 4 hours | 7.43 (15.9) | 36.3 (42.8) | 37.0 (37.5)
  After dose 5 hours: number analyzed (Participants) | 8 | 12 | 20
  After dose 5 hours | 11.6 (28.5) | 29.7 (41.9) | 44.4 (34.3)
  After dose 6 hours: number analyzed (Participants) | 7 | 11 | 18
  After dose 6 hours | 10.7 (27.0) | 32.4 (41.4) | 40.4 (35.9)
Statistical Analysis 1: Comparison: Dronabinol vs Vaporized Cannabis 3.7% THC/5.6% CBD; Test type: Superiority; p = 0.24, Regression, Linear — Area under the time concentration curve (AUC) was calculated as the aggregate effect of response and compared between the arms
Statistical Analysis 2: Comparison: Placebos vs Dronabinol; Test type: Superiority; p = 0.080, Regression, Linear — [p-value comment as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Placebos vs Vaporized Cannabis 3.7% THC/5.6% CBD; Test type: Superiority; p = 0.005, Regression, Linear — [p-value comment as in outcome 9, analysis 1]

10. Secondary Outcome: Marijuana Subscale (M-scale) of the Addiction Research Center Inventory
Description: The Marijuana subscale (M-scale) of the Addiction Research Center Inventory consists of 12 true or false questions corresponding to symptoms of cannabis intoxication; the minimum and maximum scores are 0 and 12 respectively. A higher score indicates a worse score. The questions were rephrased to evaluate the experience from the past week rather than an acute response to cannabis.
Time Frame: 8 weeks
Population: There were missing values.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebos | Dronabinol | Vaporized Cannabis 3.7% THC/5.6% CBD
Number analyzed (Participants) | 37 | 36 | 42
score on a scale
  Week 1 | 1.59 (2.02) | 1.81 (1.72) | 2.31 (2.28)
  Week 3: number analyzed (Participants) | 30 | 34 | 39
  Week 3 | 1.63 (2.11) | 2.47 (2.21) | 2.33 (1.91)
  Week 5: number analyzed (Participants) | 29 | 29 | 36
  Week 5 | 1.31 (2.19) | 2.93 (2.51) | 2.67 (2.41)
  Week 7: number analyzed (Participants) | 28 | 28 | 35
  Week 7 | 1.61 (2.41) | 2.46 (2.38) | 2.80 (2.47)
  Week 8: number analyzed (Participants) | 27 | 28 | 36
  Week 8 | 1.11 (1.95) | 2.29 (2.34) | 2.31 (2.36)
Statistical Analysis 1: Comparison: Dronabinol vs Vaporized Cannabis 3.7% THC/5.6% CBD; Test type: Superiority; p = 0.60, unstructured covariance model
Statistical Analysis 2: Comparison: Placebos vs Dronabinol; Test type: Superiority; p = 0.40, unstructured covariance model
Statistical Analysis 3: Comparison: Placebos vs Vaporized Cannabis 3.7% THC/5.6% CBD; Test type: Superiority; p = 0.72, unstructured covariance model

11. Secondary Outcome: Cold Pressor Test - Pain Sensitivity
Description: Each Cold Pressure Test will begin with an immersion of the left hand into a warm water bath for 3 min. During this time, blood pressure and heart rate will be measured. After removal of the hand from the warm water, skin temperature of the thumbpad will be recorded and participants will listen to a standardized script describing the procedures. Participants will then immerse the left hand into the cold water bath, and will be instructed to report the first painful sensation after immersion. They will then be asked to tolerate the stimulus as long as possible, but will be permitted to withdraw their hand from the cold water at any point. Maximum immersion time will be 2 min. Latency to first feel pain (pain sensitivity) and latency to withdraw the hand from the water (pain tolerance) will be recorded. Blood pressure and heart rate will be measured before and after each immersion using the arm that was not immersed in the water bath.
Time Frame: 8 weeks
Population: There were missing values
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Placebos | Dronabinol | Vaporized Cannabis 3.7% THC/5.6% CBD
Number analyzed (Participants) | 37 | 33 | 37
seconds
  Pain sensitivity Baseline | 20.0 (26.5) | 18.3 (21.8) | 26.3 (30.1)
  Week 1: number analyzed (Participants) | 24 | 25 | 28
  Week 1 | 29.4 (36.9) | 23.0 (31.6) | 20.5 (29.3)
  Week 3: number analyzed (Participants) | 19 | 27 | 26
  Week 3 | 21.9 (27.5) | 18.8 (22.6) | 21.0 (23.5)
  Week 5: number analyzed (Participants) | 18 | 21 | 29
  Week 5 | 20.9 (28.4) | 20.4 (24.8) | 24.7 (28.8)
  Week 7: number analyzed (Participants) | 18 | 22 | 23
  Week 7 | 20.4 (26.6) | 21.5 (25.7) | 20.9 (24.7)
  Week 8: number analyzed (Participants) | 23 | 21 | 25
  Week 8 | 21.1 (24.3) | 15.8 (11.0) | 23.9 (30.6)
Statistical Analysis 1: Comparison: Dronabinol vs Vaporized Cannabis 3.7% THC/5.6% CBD; Test type: Superiority; p = 0.19, unstructured covariance model — The average change of pain sensitivity (weeks 5-8 at the treatment period) from baseline were compared between the arms using an unstructured covariance model
Statistical Analysis 2: Comparison: Placebos vs Dronabinol; Test type: Superiority; p = 0.70, unstructured covariance model — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Placebos vs Vaporized Cannabis 3.7% THC/5.6% CBD; Test type: Superiority; p = 0.36, unstructured covariance model — [p-value comment as in outcome 11, analysis 1]

12. Secondary Outcome: Cannabis Withdrawal Scale - Withdrawal Intensity
Description: The Cannabis Withdrawal Scale is an assessment tool used to quantify the presence and intensity of various withdrawal symptoms (e.g., strange dreams, mood swings, depression, lack of appetite, and an inability to get to sleep). Range of scores for withdrawal intensity is from 0 to 190. A higher score is a worse score.
Time Frame: Week 8 and Week 10
Population: Some subjects dropped out before completing the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebos | Dronabinol | Vaporized Cannabis 3.7% THC/5.6% CBD
Number analyzed (Participants) | 28 | 27 | 35
score on a scale
  Week 8: number analyzed (Participants) | 26 | 26 | 28
  Week 8 | 13.5 (23.7) | 6.12 (8.98) | 12.4 (25.2)
  Week 10: number analyzed (Participants) | 28 | 25 | 35
  Week 10 | 12.7 (25.1) | 6.32 (10.2) | 9.97 (20.1)
Statistical Analysis 1: Comparison: Dronabinol vs Vaporized Cannabis 3.7% THC/5.6% CBD; Change in withdrawal intensity from week 8 to week 10 was compared between the two arms; Test type: Superiority; p = .14, Regression, Linear
Statistical Analysis 2: Comparison: Placebos vs Dronabinol; Change in withdrawal intensity from week 8 to week 10 was compared between the two arms; Test type: Superiority; p = .60, Regression, Linear
Statistical Analysis 3: Comparison: Placebos vs Vaporized Cannabis 3.7% THC/5.6% CBD; Change in withdrawal intensity from week 8 to week 10 was compared between the two arms; Test type: Superiority; p = .34, Regression, Linear

13. Secondary Outcome: Driving Simulation (Lane Tracking)
Description: Lane Tracking: This task requires subjects to drive down a straight 2-lane road, maintain a constant speed of 55 mph, maintain appropriate lane position, and respond to divided attention tasks in the upper corners of the screen. The primary outcome is standard deviation of lateral deviation (swerving) with a score range of 0.51 - 3.24. A higher score indicates worse performance.
  The driving simulation assessments are conducted in a substudy, which only includes completers with a valid driver's license and who agreed to participate in the substudy.
Time Frame: 270 minutes
Population: There are some missing values
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebos | Dronabinol | Vaporized Cannabis 3.7% THC/5.6% CBD
Number analyzed (Participants) | 5 | 11 | 16
score on a scale
  Pre Dose | 0.75 (0.18) | 1.28 (0.65) | 1.14 (0.41)
  After First Dose 30 minutes | 1.18 (0.43) | 1.41 (0.61) | 1.12 (0.32)
  After First Dose 100 minutes | 1.12 (0.57) | 1.78 (0.87) | 1.21 (0.35)
  After First Dose 230 minutes | 1.31 (0.57) | 1.51 (0.76) | 1.11 (0.25)
  After Second Dose 30 minutes | 1.13 (0.47) | 1.65 (0.79) | 1.24 (0.39)
Statistical Analysis 1: Comparison: Dronabinol vs Vaporized Cannabis 3.7% THC/5.6% CBD; Test type: Superiority; p = 0.34, unstructured covariance model
Statistical Analysis 2: Comparison: Placebos vs Vaporized Cannabis 3.7% THC/5.6% CBD; Test type: Superiority; p = 0.007, unstructured covariance model
Statistical Analysis 3: Comparison: Placebos vs Dronabinol; Test type: Superiority; p = 0.055, unstructured covariance model

14. Secondary Outcome: Driving Simulation (Car Following)
Description: Car Following: This simulation examines the participant's ability to closely match the speed of an automobile in front of them. Participants are to follow a lead vehicle at a safe and constant distance. The primary outcome is coherence between the participant and lead cars (a general correlation [0-1] of the participant's ability to accurately track the speed variations of the lead car. A higher score indicates worse performance.
  The driving simulation assessments are conducted in a substudy, which only includes completers with a valid driver's license and who agreed to participate in the substudy.
Time Frame: 270 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebos | Dronabinol | Vaporized Cannabis 3.7% THC/5.6% CBD
Number analyzed (Participants) | 5 | 11 | 16
score on a scale
  Pre Dose | 0.70 (0.17) | 0.62 (0.20) | 0.49 (0.29)
  After First Dose 30 minutes | 0.75 (0.13) | 0.71 (0.20) | 0.61 (0.23)
  After First Dose 100 minutes | 0.59 (0.33) | 0.68 (0.20) | 0.56 (0.22)
  After First Dose 230 minutes | 0.72 (0.24) | 0.60 (0.27) | 0.62 (0.25)
  After Second Dose 30 minutes | 0.74 (0.19) | 0.68 (0.26) | 0.60 (0.22)
Statistical Analysis 1: Comparison: Dronabinol vs Vaporized Cannabis 3.7% THC/5.6% CBD; Test type: Superiority; p = 0.69, unstructured covariance model
Statistical Analysis 2: Comparison: Placebos vs Vaporized Cannabis 3.7% THC/5.6% CBD; Test type: Superiority; p = 0.79, unstructured covariance model
Statistical Analysis 3: Comparison: Placebos vs Dronabinol; Test type: Superiority; p = 0.97, unstructured covariance model

15. Secondary Outcome: Locally Developed Psychoactive Effect Scale - High
Description: A total of 15 separate VAS ratings will be presented as a 100-mm horizontal line, anchored on the left with 'not at all' and on the right with 'extremely'. Participants will pencil in a vertical line along the horizontal line that represents their current feeling (questions usually phrased, 'During the past week, did you feel ___after consuming the vaporized cannabis?'). Ratings will be: any drug effect, a good drug effect, a bad drug effect, high, drunk, impaired, stoned, as if you liked the drug effect, sedated, confused, nauseous, like you desired more of the drug, anxious, down, and very hungry.
  This is a substudy. Drug "high" will be presented. Range of scores is from 0 to 100. A higher score is a worse score.
Time Frame: 6 hours
Population: There are some missing values
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebos | Dronabinol | Vaporized Cannabis 3.7% THC/5.6% CBD
Number analyzed (Participants) | 8 | 13 | 21
score on a scale
  After dose 1 hour: number analyzed (Participants) | 8 | 13 | 20
  After dose 1 hour | 5.38 (12.2) | 14.9 (31.5) | 49.8 (30.7)
  After dose 2 hours | 5.75 (14.7) | 25.8 (38.1) | 36.7 (27.1)
  After dose 3 hours: number analyzed (Participants) | 8 | 12 | 21
  After dose 3 hours | 5.56 (13.2) | 31.8 (40.5) | 20.5 (22.5)
  After dose 4 hours: number analyzed (Participants) | 7 | 13 | 21
  After dose 4 hours | 4.00 (7.00) | 28.6 (32.5) | 29.5 (32.8)
  After dose 5 hours: number analyzed (Participants) | 8 | 12 | 20
  After dose 5 hours | 1.75 (1.83) | 21.5 (36.9) | 43.9 (32.8)
  After dose 6 hours: number analyzed (Participants) | 7 | 11 | 18
  After dose 6 hours | 1.71 (3.40) | 24.8 (38.7) | 31.7 (30.3)
Statistical Analysis 1: Comparison: Dronabinol vs Vaporized Cannabis 3.7% THC/5.6% CBD; Test type: Superiority; p = 0.21, Regression, Linear — [p-value comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: Placebos vs Dronabinol; Test type: Superiority; p = 0.029, Regression, Linear — [p-value comment as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Placebos vs Vaporized Cannabis 3.7% THC/5.6% CBD; Test type: Superiority; p = 0.001, Regression, Linear — [p-value comment as in outcome 9, analysis 1]

16. Secondary Outcome: Cannabis Withdrawal Scale - Negative Impact of Withdrawal
Description: The Cannabis Withdrawal Scale is an assessment tool used to quantify the presence and intensity of various withdrawal symptoms (e.g., strange dreams, mood swings, depression, lack of appetite, and an inability to get to sleep). The outcome is measured during the tapering period (weeks 8 and 10), at which patients slowly withdrew from medication over two weeks. Range of scores for the negative impact of withdrawal is from 0 to 190. A higher score is a worse score.
Time Frame: Week 8, Week 10
Population: Some subjects dropped out before completing the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebos | Dronabinol | Vaporized Cannabis 3.7% THC/5.6% CBD
Number analyzed (Participants) | 28 | 27 | 35
score on a scale
  Week 8: number analyzed (Participants) | 26 | 26 | 28
  Week 8 | 8.42 (22.9) | 3.42 (7.22) | 10.3 (24.6)
  Week 10: number analyzed (Participants) | 28 | 25 | 35
  Week 10 | 8.18 (24.0) | 2.32 (8.63) | 4.31 (10.5)
Statistical Analysis 1: Comparison: Dronabinol vs Vaporized Cannabis 3.7% THC/5.6% CBD; Change in negative impact of withdrawal from week 8 to week 10 was compared between the two arms; Test type: Superiority; p = 0.084, Regression, Linear
Statistical Analysis 2: Comparison: Placebos vs Dronabinol; Change in negative impact of withdrawal from week 8 to week 10 was compared between the two arms; Test type: Superiority; p = 0.98, Regression, Linear
Statistical Analysis 3: Comparison: Placebos vs Vaporized Cannabis 3.7% THC/5.6% CBD; Change in negative impact of withdrawal from week 8 to week 10 was compared between the two arms; Test type: Superiority; p = 0.085, Regression, Linear

17. Secondary Outcome: Cold Pressor Test - Pain Tolerance
Description: as for outcome 11
Time Frame: 8 weeks
Population: There were some missing values
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Placebos | Dronabinol | Vaporized Cannabis 3.7% THC/5.6% CBD
Number analyzed (Participants) | 37 | 33 | 37
seconds
  Baseline | 47.2 (42.0) | 40.6 (34.1) | 58.3 (46.0)
  Week 1: number analyzed (Participants) | 24 | 25 | 28
  Week 1 | 50.5 (40.4) | 44.8 (46.9) | 60.9 (48.8)
  Week 3: number analyzed (Participants) | 19 | 27 | 26
  Week 3 | 46.2 (38.0) | 40.0 (34.3) | 64.3 (49.3)
  Week 5: number analyzed (Participants) | 18 | 21 | 29
  Week 5 | 41.4 (39.5) | 43.6 (41.5) | 60.7 (45.9)
  Week 7: number analyzed (Participants) | 18 | 22 | 23
  Week 7 | 61.7 (53.8) | 44.2 (40.4) | 54.7 (42.9)
  Week 8: number analyzed (Participants) | 23 | 21 | 25
  Week 8 | 37.9 (35.0) | 37.5 (32.4) | 62.3 (45.8)
Statistical Analysis 1: Comparison: Dronabinol vs Vaporized Cannabis 3.7% THC/5.6% CBD; Test type: Superiority; p = 0.95, unstructured covariance model — The average change of pain tolerance (weeks 5-8 at the treatment period) from baseline were compared between the arms using an unstructured covariance model
Statistical Analysis 2: Comparison: Placebos vs Dronabinol; Test type: Superiority; p = 0.78, unstructured covariance model — [p-value comment as in outcome 17, analysis 1]
Statistical Analysis 3: Comparison: Placebos vs Vaporized Cannabis 3.7% THC/5.6% CBD; Test type: Superiority; p = 0.99, unstructured covariance model — [p-value comment as in outcome 17, analysis 1]

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Placebos | Dronabinol | Vaporized Cannabis 3.7% THC/5.6% CBD
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/43 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/43 | 0/44
Other Adverse Events (participants affected / at risk) | 30/44 | 31/43 | 30/44
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebos (N=44) | Dronabinol (N=43) | Vaporized Cannabis 3.7% THC/5.6% CBD (N=44)
Nausea (Gastrointestinal disorders) | 8 (10) | 11 (12) | 11 (14)
Confusion (Nervous system disorders) | 8 (10) | 10 (14) | 7 (9)
Lethargy (Nervous system disorders) | 19 (25) | 16 (32) | 23 (37)
Dry Mouth (Nervous system disorders) | 8 (9) | 19 (26) | 12 (17)
Headache (Nervous system disorders) | 14 (18) | 12 (12) | 14 (21)
Abnormal cognition (Nervous system disorders) | 3 (3) | 10 (12) | 10 (13)
Depression (Nervous system disorders) | 9 (10) | 8 (10) | 6 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 8 (9) | 11 (14)
Vomiting (Nervous system disorders) | 2 (3) | 4 (4) | 6 (6)
Dizzy (Nervous system disorders) | 7 (8) | 7 (8) | 9 (9)
Emotional Changes (Nervous system disorders) | 10 (10) | 9 (13) | 14 (15)
Sleeping Problems (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paranoia (Nervous system disorders) | 2 (4) | 6 (7) | 2 (3)
Stomach Pain (General disorders) | 2 (2) | 6 (8) | 5 (6)
Abnormal Coordination (Nervous system disorders) | 6 (6) | 10 (15) | 8 (10)
Anxiety (Nervous system disorders) | 8 (8) | 7 (10) | 8 (10)
Back/Flank Paresthesia (Nervous system disorders) | 4 (4) | 6 (8) | 6 (7)
Abnormal Dreams (Nervous system disorders) | 5 (7) | 3 (5) | 8 (13)
Back/Flank Numbness (Nervous system disorders) | 6 (6) | 1 (1) | 3 (3)
Abnormal Balance (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Orthostatic Hypotension (Nervous system disorders) | 3 (4) | 1 (2) | 2 (2)
Abnormal heart rate (Nervous system disorders) | 2 (4) | 2 (2) | 4 (4)
Vision Alteration (Nervous system disorders) | 2 (2) | 3 (3) | 2 (2)
Blood pressure decreased (Nervous system disorders) | 1 (1) | 2 (3) | 1 (1)
Abdomen/Groin/Pelvis Pain (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2)
Blood pressure increased (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Face/Jaw/Lips dry (General disorders) | 0 (0) | 1 (1) | 1 (1)
Generalized/Multiple site numbness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Behavior changes (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Bronchial washing nausea (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Cronic bronchitis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Sexual drive alteration (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-10-10): https://cdn.clinicaltrials.gov/large-docs/92/NCT02460692/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-24): https://cdn.clinicaltrials.gov/large-docs/92/NCT02460692/SAP_001.pdf